CLINICAL TRIAL: NCT04979052
Title: Safety and Efficacy of Recombinant Interferon-Gamma 1b (rIFN-Gamma 1b) Given With Standard Therapy in Patients With Candidemia
Brief Title: Safety and Efficacy of Interferon-Gamma 1b in Patients With Candidemia
Acronym: HDM-FUN Cand
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDM-FUN-Candidemia
Record Dates: First submitted 2020-11-09; First posted 2021-07-27 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Candidemia
Keywords: Interferon Gamma 1b
MeSH Terms: conditions — Candidemia | interventions — interferon gamma-1b

STUDY DESIGN:
Intervention Model Description: Open label adaptive randomized interventional study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Interferon-Gamma (Active Comparator): Recombinant Interferon-Gamma 1b combined with standard therapy
  Interventions: Drug: Interferon Gamma-1B
- Standard of care (No Intervention): Standard of care antifungal therapy according tot ESCMID/EFISG (Europe) or ISDA (US) guidelines.

INTERVENTIONS:
Drug: Interferon Gamma-1B — 100 microgram per day, three times a week, subcutaneous. The duration of the treatment is twelve days or until hospital discharge.
  Other Names: Immukin
  Arms: Interferon-Gamma

SUMMARY:
A multi-center open label adaptive randomized interventional phase 2 study to evaluate safety and efficacy of rIFN-y treatment in patiens with candidemia.

DETAILED DESCRIPTION:
A multi-center open label adaptive randomized interventional phase 2 study to evaluate safety and efficacy of rIFN-y treatment in patiens with candidemia. Patients will be randomized 1:1 between intervention (rIFN-y immunotherapy, subcutaneous dose of 100miicrogram thrice weekly for two weeks or until hospital discharge) in addition to standard of care versus controls (standard of care). Standard of care antifungal therapy is according to ESCMID/EFISG (Europe) or IDSA (US) guidelines. We will assess the effect on clinical outcome and investigate relevant biomarkers that can guide this immunotherapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females (who must agree to use barrier methods of contraception during the study therapy period, women of childbearing age must have a negative urine pregnancy or serum test at baseline).
* Subjects who are 18 years of age or older.
* Subjects with at least one positive blood culture isolation of Candida species from a specimen drawn within 120 hours prior to study entry.
* Subjects who have clinical evidence of infection sometime within 120 hours prior to enrolment, including at least one of the following:

  * Temperature >37.8 ˚C on two occasions at least four hours apart or one measurement > 38.2 ˚C
  * Systolic blood pressure <90 or a >30 mmHg decrease in systolic blood pressure from the subject's normal baseline or the need for vassopressive therapy.
  * Signs of inflammation (swelling, heat, erythema, purulent drainage) from a site infected with Candida (e.g. joint, skin, eye, bone, oesophagus).
  * Radiologic findings of invasive candidiasis.
* Subject or their legal representative must sign a written informed consent form.
* In case a patient eligible to participate in this study is incapacitated and as such unable to personally provide informed consent, a written consent form must be signed by their legal representative.

  * Only incapacitated patients that can be expected to regain the capability to consent will be included in this study. In this case, informed consent will be discussed personally with the study participant after recovery.
  * The inclusion of incapacitated subjects will only be performed under the above conditions in a country in which such an approach is legal and deemed ethically acceptable.

Exclusion Criteria:

* Subjects with a history of allergy or intolerance to rIFN-γ,or any other IMP ingredient or with a history of immediate type hypersensitivity to latex/rubber.
* Subjects with a history of documented epileptic seizures.
* Subjects with severe liver failure ((>5x upper limit AST or ALT or impaired synthesis of proteins such as coagulation factors manifested by increased prothrombin time).
* Treatment with heterologous serum proteins, or immunological preparations such as vaccines, toxins, serums and allergens within three days before trial enrolment.
* Women who are pregnant or lactating.
* Subjects who are unlikely to survive more than 24 hours.
* Subjects who have failed previous systemic antifungal therapy for the Candida spp.

infection which is being studied.

* Subjects who have received more than 120 hours of systemic antifungal therapy for the current episode, within 120 hours prior to study entry.
* With respect to incapacitated subjects:
* Any patient that is deemed incapable of personally providing informed consent due to a neurodegenerative disease, genetic syndrome, and/or perinatal asphyxia, will not be eligible for inclusion in this trial.
* Any incapacitated subject that is not expected to recover to a point where they will personally be able to provide informed consent will not be eligible for inclusion in this trial. Patients with renal failure or dialysis do not have a contraindication for treatment with rIFN-y and can be included in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to first negative blood culture | Day 14

SECONDARY OUTCOMES:
Time to treatment success | Day 14
  microbiological eradication of Candida from the blood and any other site of infection; resolution of fever; resolution of other diagnostic variables, such as imaging results, where applicable; and no new signs of infection. The time at which all the variables are met is defined as the date of resolution of infection.
Percentage of patients with mycological outcomes | through intervention completion, an average at day 11 and 2 and 4 weeks after intervention completion
Percentage of patients with treatment success | through intervention completion, an average at day 11 and 2 and 4 weeks after intervention completion
Overall survival | Study day 28
Number of patients with Treatment Emergent Adverse Events (TEAEs). | Study day 49
Sequential Organ Failure Assessment (SOFA) score | Study day 14
Adverse events | Study day 14
Body weight | Study day 49
  kg
BMI | Study day 49
  kg/m^2
Prealbumin | Study day 49
  mg/dl
Total lymphocytes | Study day 49
  10^9/L
Cholesterol | Study day 49
  mmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Frank vd Veerdonk, Dr., Principal Investigator — Radboud University Medical Center
Locations (6):
- Duke University, Durham, North Carolina, United States
- Klinikum Der Johann Wolfgang Von Goethe Universitaet, Frankfurt am Main, Germany
- Hellenic Institute for the Study of Sepsis (HISS), Athens, Greece
- Radboudumc, Nijmegen, Gelderland, Netherlands
- Universitatea de Medicina si Farmacie luliu Hatieganu, Cluj-Napoca, Romania
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No